CLINICAL TRIAL: NCT00902577
Title: Multicenter, Phase II Assessment of Tumor Hypoxia in Glioblastoma Using 18F-Fluoromisonidazole (FMISO) With PET and MRI
Brief Title: MRI and PET/FMISO In Assessing Tumor Hypoxia in Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2011-01912; NCI-2011-01912 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000640413 (Registry Identifier: ClinicalTrials.gov); ACRIN 6684 (Other: American College of Radiology Imaging Network); ACRIN-6684 (Other: CTEP); U01CA080098 (NIH)
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-03

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — fluoromisonidazole; Magnetic Resonance Spectroscopy; X-Rays

ARMS (1):
- Diagnostic (MRI and PET using FMISO) (Experimental): Two weeks before initiation of chemoradiotherapy with temozolomide, patients undergo MRI (DSC, DCE,DWI and MRS) and PET scan using FMISO. A subset of 15 patients undergo FMISO PET scans approximately 1 week before chemoradiotherapy.
  Interventions: Drug: FMISO; Other: MRI; Other: PET; Other: MRS

INTERVENTIONS:
Drug: FMISO — FMISO PET scans
  Other Names: 18F-fluoromisonidazole; 18F-MISO; 18F-Misonidazole
Other: MRI — Undergo MRI
  Other Names: Magnetic Resonance Imaging (MRI); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance; MRI Scan; NMR Imaging; Nuclear Magnetic Resonance Imaging (NMRI); Nuclear Magnetic Resonance Imaging; Medical Imaging, Nuclear Magnetic Resonance; Magnetic Resonance (MR)
Other: PET — Undergo FMISO PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET Scan; Positron Emission Tomography; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Other: MRS
  Other Names: Magnetic Resonance Spectroscopy (MRS); Magnetic Resonance Imaging Spectroscopy (MRIS); Magnetic Resonance Spectroscopy Imaging (MRSI)

SUMMARY:
This phase II trial is studying how well positron emission tomography (PET) scan using 18F-fluoromisonidazole works when given together with magnetic resonance imaging (MRI) ) in assessing tumor hypoxia in patients with newly diagnosed glioblastoma multiforme (GBM). Diagnostic procedures, such as MRI and PET scan using 18F-fluoromisonidazole (FMISO), may help predict the response of the tumor to the treatment and allow doctors to plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the association of baseline FMISO PET uptake (hypoxic volume [HV]), highest tumor:blood ratio [T/Bmax]) and MRI parameters (Ktrans, CBV) with overall survival (OS) in participants with newly diagnosed GBM.

SECONDARY OBJECTIVES:

I. To determine the association of baseline FMISO PET uptake (HV, T/Bmax) and MRI parameters (Ktrans, CBV) with time to progression (TTP) and 6-month progression free survival (PFS-6) in participants with newly diagnosed GBM.

II. To assess the reproducibility of the baseline FMISO PET uptake parameters by implementing baseline "test" and "retest" PET scans (performed within 1 to 7 days of each other).

III. To assess the correlation between highest tissue:cerebellum ratio [T/Cmax] and T/Bmax at baseline.

IV. To assess the correlation between other MRI parameters (for example Gadolinium-enhanced T1-weighted (T1Gd), vessel caliber index (VCI), , CBV-S, apparent diffusion coefficient (ADC) , N-acetylaspartate (NAA) to choline (Cho) ratio, blood oxygenation level-dependent (BOLD), T2) and OS, TTP, and PFS-6.

OUTLINE: This is a multicenter study.

Two weeks before initiation of chemoradiotherapy with temozolomide, patients undergo MRI and PET scan using FMISO. A subset of 15 patients undergo FMISO PET scans approximately 1 week before chemoradiotherapy. Blood samples are collected at baseline and periodically during study to compare image measures of tissue uptake of FMISO to blood concentrations. Tumor samples are collected from diagnostic biopsy or surgery for analysis of tumor hypoxic markers and methylguanine methyl transferase by immunohistochemical and Polymerase chain reaction (PCR) assays.

After completion of study therapy, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* Newly diagnosed glioblastoma multiforme (GBM), World Health Organization (WHO) grade IV based on pathology confirmation
* Residual tumor after surgery (amount of residual tumor will not impact patient eligibility and visible residual disease can include T2/FLAIR hyperintensity)

  * Note: If patient had a biopsy only, postoperative MRI is not needed to assess residual tumor prior to enrollment
* Scheduled to receive standard fractionated radiation therapy
* Scheduled to receive Temozolomide (TMZ) in addition to radiation therapy
* Karnofsky Performance Score > 60

Exclusion Criteria:

* Pregnant or breastfeeding (if a female is of child-bearing potential, and unsure of pregnancy status, a standard urine pregnancy test should be done)
* Scheduled to receive chemotherapy, immunotherapy, or investigational agents in trials unwilling to share data with ACRIN (i.e., additional therapy added to radiation and TMZ is allowed if ACRIN is able to obtain treatment information)
* Not suitable to undergo MRI or use the contrast agent Gd because of:
* Claustrophobia
* Presence of metallic objects or implanted medical devices in body (i.e., cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
* Sickle cell disease
* Renal failure
* Reduced renal function, as determined by Glomerular Filtration Rate (GFR) < 30 mL/min/1.73 m^2 based on a serum creatinine level obtained within 28 days prior to registration
* Presence of any other co-existing condition which, in the judgment of the investigator, might increase the risk to the subject
* Presence of serious systemic illness, including: uncontrolled intercurrent infection, uncontrolled malignancy, significant renal disease, or psychiatric/social situations which might impact the survival endpoint of the study or limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to FMISO; an allergic reaction to nitroimidazoles is highly unlikely
* Not suitable to undergo PET or MRI, including weight greater than 350 lbs (the weight limit for the MRI and PET table)
* Prior treatment with implanted radiotherapy or chemotherapy sources such as wafers of polifeprosan 20 with carmustine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08-24 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, Principal Investigator — American College of Radiology Imaging Network
Locations (14):
- United States (14):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - American College of Radiology Imaging Network, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Ratai EM, Zhang Z, Fink J, Muzi M, Hanna L, Greco E, Richards T, Kim D, Andronesi OC, Mintz A, Kostakoglu L, Prah M, Ellingson B, Schmainda K, Sorensen G, Barboriak D, Mankoff D, Gerstner ER; ACRIN 6684 trial group. ACRIN 6684: Multicenter, phase II assessment of tumor hypoxia in newly diagnosed glioblastoma using magnetic resonance spectroscopy. PLoS One. 2018 Jun 14;13(6):e0198548. doi: 10.1371/journal.pone.0198548. eCollection 2018. PMID 29902200
- [Result] Gerstner ER, Zhang Z, Fink JR, Muzi M, Hanna L, Greco E, Prah M, Schmainda KM, Mintz A, Kostakoglu L, Eikman EA, Ellingson BM, Ratai EM, Sorensen AG, Barboriak DP, Mankoff DA; ACRIN 6684 Trial Group. ACRIN 6684: Assessment of Tumor Hypoxia in Newly Diagnosed Glioblastoma Using 18F-FMISO PET and MRI. Clin Cancer Res. 2016 Oct 15;22(20):5079-5086. doi: 10.1158/1078-0432.CCR-15-2529. Epub 2016 May 16. PMID 27185374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty patients with newly diagnosed GBM were enrolled from 11 academic centers in the United States.
Pre-assignment Details: All participants were scheduled to receive both FMISO and MRI (DCE, DSC, DWI, MRS) imaging two weeks before initiation of chemoradiotherapy with temozolomide
Groups:
- Newly Diagnosed Glioblastoma Multiforme Patients: Patients with Newly diagnosed GBM scheduled to have FMISO Positron Emission Tomography (PET) two weeks before initiation of chemoradiotherapy with temozolomide, with diagnostic DCE/DSE/DWI MRI
Period: Overall Study
Arm/Group | Newly Diagnosed Glioblastoma Multiforme Patients
Started | 50
FMISO/PET (3 images lost/Not Acquired 1 Image uninterpretable) | 38
DCE MRI (2 images lost/Not Acquired 9 Image uninterpretable) | 31
DSE MRI (2 images lost/Not Acquired 3 Image uninterpretable) | 37
DWI MRI (3 images lost/Not Acquired) | 39
Completed | 42
Not Completed | 8
Not completed — Withdrawal by Subject | 6
Not completed — FMISO production failure | 2

BASELINE CHARACTERISTICS:
Population: Patients with newly diagnosed GBM who received both FMISO-PRT imaging two weeks before initiation of chemoradiotherapy with temozolomide
Groups:
- Newly Diagnosed Glioblastoma Multiforme Patients: 42 eligible, consented patients with newly diagnosed GBM who received both FMISO-PRT and MRI imaging two weeks before initiation of chemoradiotherapy with temozolomide
Arm/Group | Newly Diagnosed Glioblastoma Multiforme Patients
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Median Tumor Volume [Median (Inter-Quartile Range); unit: mm^3] | 14.94 [.84 to 59.5]

OUTCOME MEASURES:

1. Primary Outcome: Association of Baseline FMISO PET and MRI Features With OS as Assessed Using Cox-regression Model
Description: Overall Survival (OS) was evaluated every 3 months through end of the study (up to 5 years). A variety of continuous quantitative (functional) imaging features measuring abnormal tumor vasculature (MRI) and hypoxia (FMISO) were evaluated at baseline for their association with Survival time.
  Features include
  PET Hypoxia measures:
  Peak standardized uptake values (SUVpeak); maximum tumor:blood ratio (T/Bmax); and Hypoxia Volume (HV)
  DCE MRI perfusion measures:
  Mean/median volume transfer constant for gadolinium between blood plasma and the tissue extravascular extracellular space (ktrans)
  DSC MRI tumor vasculature:
  Normalized Relative cerebral blood volume (nRCBV); and Cerebral blood flow (CBF)
  DWI MRI magnitude of diffusion of water through tissue (cell density):
  Apparent diffusion coefficient (ADC) using low and high Gaussian distributions
Time Frame: "assessed from baseline up to 5 years, survival status at 1-year reported
Population: FMISO-PET identifies the primary analysis population containing participants with interpretable FMISO images.The Evaluable study population consisted of enrolled GBM patients having an FMISO-PET procedure. Additional groups include functional MRI, with available/interpretable images.
Measure: Count of Participants; unit: Participants
Groups:
- Evaluable: 42 participants with imaging (FMISO-PET, DCE/DSC/DWI MRI)
- FMISO-PET: Quantitative PET measurements Hypoxic Volume (HV) Max tumor:blood ratio (TBmax) Peak Standardized uptake Values (SUVpeak)
- DSC MRI: Quantitative DSC measurements:
  Normalized rCBV [Relative cerebral blood volume] Normalized rCBF[Relative cerebral blood flow]
- DCE MRI: Quantitative DCE measurements Mean vascular permeability (ktrans) Median Ktrans
- DWI-MRI: Apparent diffusion coefficient (ADC) Low and High
Arm/Group | Evaluable | FMISO-PET | DSC MRI | DCE MRI | DWI-MRI
Number analyzed (Participants) | 42 | 38 | 37 | 31 | 39
Participants
  OS-1 Alive | 25 | 22 | 24 | 20 | 24
  OS-1 Death | 17 | 16 | 13 | 11 | 15
Statistical Analysis 1: Comparison: FMISO-PET; FMISO selectively binds to hypoxic tissues so that SUVpeak within a region provides a measure of tumor hypoxia.: This marker was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.048, Regression, Cox; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [1.0 to 2.36]
Statistical Analysis 2: Comparison: FMISO-PET; T/Bmax is the pixel in the tumor region with the maximum tumor:blood ratio (T/Bmax) and T/Bmax depicts the magnitude of the hypoxia TBmax was modeled with a univariate Cox regression model for OS time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported. The study was designed to enroll 46 evaluable participants to detect a log hazard ratio of 1.279 for TBmax with HV as a covariate with a 50% event rate; Test type: Other; p = 0.50, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [.75 to 1.81]
Statistical Analysis 3: Comparison: FMISO-PET; Hypoxia Volume (HV) depicts the volume of tumor that has crossed the threshold for hypoxia. Hypoxic Volume (HV) was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.90, Regression, Cox; Hazard Ratio (HR) = 1.00, 0.97% CI 2-sided [0.97 to 1.03]
Statistical Analysis 4: Comparison: DCE MRI; ktrans reflects the rate of gadolinium moves from plasma to extravascular extracellular space (predominantly though blood flow and capillary leakage). Mean ktrans were computed using a matrix-based linearization method to fit tissue ∆R1(t) to the extended Tofts model Mean ktrans was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.024, Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [1.02 to 1.34] — HR reported per 0.01 increase
Statistical Analysis 5: Comparison: DCE MRI; ktrans reflects the rate of gadolinium moves from plasma to extravascular extracellular space (predominantly though blood flow and capillary leakage). Median ktrans were computed using a matrix-based linearization method to fit tissue ∆R1(t) to the extended Tofts model. Median ktrans was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.045, Regression, Cox; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.01 to 1.72] — HR reported per 0.01 increase
Statistical Analysis 6: Comparison: DSC MRI; Relative cerebral blood volume (RCBV) maps, computed from the integral of ∆R2*(t), were corrected for leakage effects and normalized to normal appearing white matter (nRCBV); nRCBV provides a measure of tumor vasculature and was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.31, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.90 to 1.37]
Statistical Analysis 7: Comparison: DSC MRI; cerebral blood flow (CBF) maps were was normalized to the mean of the region of interest (ROI) in normal appearing white matter to produce the nCBF and provide another measure of vascular permeability and perfusion nCBF was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.51, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.88 to 1.29]
Statistical Analysis 8: Comparison: DWI-MRI; Apparent Diffusion Coefficient (ADC) measures water diffusion through tissue. Cerebral infarction leads to diffusion restriction resulting in a low ADC signal in the infarcted area. A double Gaussian mixed model was fit to the ADC histogram and the mean of the lower ADC curve, was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.9700, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.79 to 1.26]
Statistical Analysis 9: Comparison: DWI-MRI; Apparent Diffusion Coefficient (ADC) measures water diffusion through tissue. Cerebral infarction leads to diffusion restriction resulting in a low ADC signal in the infarcted area. A double Gaussian mixed model was fit to the ADC histogram and the mean of the higher ADC curve, was modeled with a univariate Cox regression model for overall survival (OS) time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.9007, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.91 to 1.09]

2. Secondary Outcome: Association of Baseline FMISO PET and MRI Features With Time-to-Progression (TTP)
Description: Disease progression was defined by Macdonald criteria. PFS was evaluated every 3months through the end of study (up to 5yrs), features were measured at baseline.
  Quantitative imaging features measuring abnormal tumor vasculature (MRI) and hypoxia (FMISO) were evaluated for their association with TTP (cox model) and to discriminate between responders and non-responders at 6 and 9 mos (PFS6 and PFS9) (logistic) Features include
  PET Hypoxia measures:
  Peak standardized uptake values (SUVpeak); maximum tumor:blood ratio (T/Bmax); and Hypoxia Volume (HV)
  DCE MRI perfusion measures:
  Mean/median volume transfer constant for gadolinium between blood plasma and the tissue extravascular extracellular space (ktrans)
  DSC MRI tumor vasculature:
  Normalized Relative cerebral blood volume (nRCBV); and Cerebral blood flow (CBF)
  DWI MRI magnitude of diffusion of water through tissue (cell density):
  Apparent diffusion coefficient (ADC) using low and high Gaussian distributions
Time Frame: assessed from baseline up to 5 years, progression status at months 6 and 9 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluable | FMISO-PET | DSC MRI | DCE MRI | DWI-MRI
Number analyzed (Participants) | 42 | 38 | 37 | 31 | 39
Participants
  6 month Progression Status: Progression Free | 29 | 26 | 27 | 20 | 28
  6 month Progression Status: Progressed | 13 | 12 | 10 | 11 | 11
  9 Month Progression Status: Progression Free | 19 | 17 | 18 | 12 | 18
  9 Month Progression Status: Progressed | 23 | 21 | 19 | 19 | 21
Statistical Analysis 1: Comparison: FMISO-PET; FMISO selectively binds to hypoxic tissues so that SUVpeak within a region provides a measure of tumor hypoxia. This marker was modeled with a univariate Cox regression model for Progression Free Survival time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.33, Regression, Cox; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [.80 to 1.91]
Statistical Analysis 2: Comparison: FMISO-PET; T/Bmax is the pixel in the tumor region with the maximum tumor:blood ratio (T/Bmax) and T/Bmax depicts the magnitude of the hypoxia TBmax was modeled with a univariate Cox regression model for PFS time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.72, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [.61 to 1.4]
Statistical Analysis 3: Comparison: FMISO-PET; Hypoxia Volume (HV) depicts the volume of tumor that has crossed the threshold for hypoxia. Hypoxic Volume (HV) was modeled with a univariate Cox regression model for PFS time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.355, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [.98 to 1.04]
Statistical Analysis 4: Comparison: DCE MRI; ktrans reflects the rate of gadolinium moves from plasma to extravascular extracellular space (predominantly though blood flow and capillary leakage). Mean ktrans were computed using a matrix-based linearization method to fit tissue ∆R1(t) to the extended Tofts model. Mean ktrans was modeled with a univariate Cox regression model for PFS time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.074, Regression, Cox; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.99 to 1.23]
Statistical Analysis 5: Comparison: DCE MRI; ktrans reflects the rate of gadolinium moves from plasma to extravascular extracellular space (predominantly though blood flow and capillary leakage). Median ktrans were computed using a matrix-based linearization method to fit tissue ∆R1(t) to the extended Tofts model. Median ktrans was modeled with a univariate Cox regression model for PFS time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.021, Regression, Cox; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [1.04 to 1.63]
Statistical Analysis 6: Comparison: DSC MRI; Relative cerebral blood volume (RCBV) maps, computed from the integral of ∆R2*(t), were corrected for leakage effects and normalized to normal appearing white matter (nRCBV); nRCBV provides a measure of tumor vasculature and was modeled with a univariate Cox regression model for PFS time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.0096, Regression, Cox; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [1.06 to 1.54]
Statistical Analysis 7: Comparison: DSC MRI; cerebral blood flow (CBF) maps were was normalized to the mean of the region of interest (ROI) in normal appearing white matter to produce the nCBF and provide another measure of vascular permeability and perfusion. nCBF was modeled with a univariate Cox regression model for PFS time. The hazard ratio, along with its 95% confidence interval and the p-value based on Wald's statistic are reported; Test type: Other; p = 0.038, Regression, Cox; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [1.01 to 1.38]
Statistical Analysis 8: Comparison: FMISO-PET; Logistic regression for SUVpeak to predict PFS6; Test type: Other; p = 0.3253, Regression, Logistic; Odds Ratio (OR) = 0.682, 95% CI 2-sided [0.318 to 1.463]
Statistical Analysis 9: Comparison: FMISO-PET; TBmax was modeled with a univariate logistic regression model for PFS6; Test type: Other; p = 0.9836, Regression, Logistic; Odds Ratio (OR) = 0.991, 95% CI 2-sided [0.403 to 2.434]
Statistical Analysis 10: Comparison: FMISO-PET; Hypoxic Volume (HV) was modeled with a logistic regression model for 6month progression free survival (PFS6); Test type: Other; p = 0.1566, Regression, Logistic; Odds Ratio (OR) = 0.957, 95% CI 2-sided [0.900 to 1.017]
Statistical Analysis 11: Comparison: DCE MRI; Mean ktrans were computed using a matrix-based linearization method to fit tissue ∆R1(t) to the extended Tofts model. Mean ktrans was modeled with a univariate logistic regression model for PFS6; Test type: Other; p = 0.9554, Regression, Logistic; Odds Ratio (OR) = 0.993, 95% CI 2-sided [0.775 to 1.273]
Statistical Analysis 12: Comparison: DCE MRI; Median ktrans were computed using a matrix-based linearization method to fit tissue ∆R1(t) to the extended Tofts model. Median ktrans was modeled with a univariate logistic regression model for PFS6; Test type: Other; p = 0.6941, Regression, Logistic; Odds Ratio (OR) = 0.919, 95% CI 2-sided [0.602 to 1.402]
Statistical Analysis 13: Comparison: DSC MRI; Relative cerebral blood volume (RCBV) maps were corrected for leakage effects and normalized to normal appearing white matter (nRCBV). nRCBV was modeled with a univariate logistic regression model for PFS6; Test type: Other; p = 0.1340, Regression, Logistic; Odds Ratio (OR) = 0.744, 95% CI 2-sided [0.506 to 1.095]
Statistical Analysis 14: Comparison: DSC MRI; cerebral blood flow (CBF) maps were was normalized to the mean of the region of interest (ROI) in normal appearing white matter to produce the nCBF. nCBF was modeled with a univariate logistic regression model for PFS6; Test type: Other; p = 0.2642, Regression, Logistic; Odds Ratio (OR) = 0.821, 95% CI 2-sided [0.580 to 1.161]
Statistical Analysis 15: Comparison: DWI-MRI; Apparent Diffusion Coefficient (ADC) low values were modeled with a univariate logistic regression model for PFS6; Test type: Other; p = 0.5069, Regression, Logistic; Odds Ratio (OR) = 0.855, 95% CI 2-sided [0.539 to 1.357]
Statistical Analysis 16: Comparison: DWI-MRI; Apparent Diffusion Coefficient (ADC) high values were modeled with a univariate Logistic regression model for PFS6; Test type: Other; p = 0.1921, Regression, Logistic; Odds Ratio (OR) = 0.884, 95% CI 2-sided [0.735 to 1.064]
Statistical Analysis 17: Comparison: FMISO-PET; FMISO selectively binds to hypoxic tissues so that SUVpeak within a region provides a measure of tumor hypoxia. Receiver Operating Characteristic(ROC) analysis was perform to determine the accuracy of this marker to predict PFS9; Test type: Other — An Area Under the Curve (AUC) with a lower bound of at least 0.5 is considered statistically significant; Area Under the Curve (AUC) = 0.61, 95% CI 2-sided [0.42 to 0.79]
Statistical Analysis 18: Comparison: FMISO-PET; T/Bmax is the pixel in the tumor region with the maximum tumor:blood ratio (T/Bmax) and T/Bmax depicts the magnitude of the hypoxia. Receiver Operating Characteristic(ROC) analysis was perform to determine the accuracy of this marker to predict PFS9; Test type: Other — An Area Under the Curve (AUC) with a lower bound of at least 0.5 is considered statistically significant; Area Under the Curve (AUC) = 0.59, 95% CI 2-sided [0.39 to 0.78]
Statistical Analysis 19: Comparison: FMISO-PET; Hypoxia Volume (HV) depicts the volume of tumor that has crossed the threshold for hypoxia. Receiver Operating Characteristic(ROC) analysis was perform to determine the accuracy of this marker to predict PFS9; Test type: Other — An Area Under the Curve (AUC) with a lower bound of at least 0.5 is considered statistically significant; Area Under the Curve (AUC) = 0.64, 95% CI 2-sided [0.46 to 0.83]
Statistical Analysis 20: Comparison: DCE MRI; mean ktrans reflects the rate of gadolinium moves from plasma to extravascular extracellular space (predominantly though blood flow and capillary leakage). Receiver Operating Characteristic(ROC) analysis was perform to determine the accuracy of mean ktrans to predict PFS9; Test type: Other — An Area Under the Curve (AUC) with a lower bound of at least 0.5 is considered statistically significant; Area Under the Curve (AUC) = 0.62, 95% CI 2-sided [0.42 to 0.83]
Statistical Analysis 21: Comparison: DCE MRI; Median ktrans reflects the rate of gadolinium moves from plasma to extravascular extracellular space (predominantly though blood flow and capillary leakage). Receiver Operating Characteristic(ROC) analysis was perform to determine the accuracy of Median ktrans to predict PFS9; Test type: Other — An Area Under the Curve (AUC) with a lower bound of at least 0.5 is considered statistically significant; Area Under the Curve (AUC) = 0.64, 95% CI 2-sided [0.44 to 0.84]
Statistical Analysis 22: Comparison: DSC MRI; nRCBV provides a measure of tumor vasculature Receiver Operating Characteristic(ROC) analysis was perform to determine the accuracy of this marker to predict PFS9; Test type: Other — An Area Under the Curve (AUC) with a lower bound of at least 0.5 is considered statistically significant; Area Under the Curve (AUC) = 0.72, 95% CI 2-sided [0.54 to 0.89]
Statistical Analysis 23: Comparison: DSC MRI; nCBF provides a measure of vascular permeability and perfusion. Receiver Operating Characteristic(ROC) analysis was perform to determine the accuracy of this marker to predict PFS9; Test type: Other — An Area Under the Curve (AUC) with a lower bound of at least 0.5 is considered statistically significant; Area Under the Curve (AUC) = 0.72, 95% CI 2-sided [0.55 to 0.89]

3. Secondary Outcome: Reproducibility of the Baseline FMISO PET Uptake Parameters as Assessed by Baseline "Test" and "Retest" PET Scans
Description: Reproducibility, defined as the variation of repeated measurements in an experiment performed under the same conditions, will be measured as the within subject coefficient of variation with upper an lower repeatability coefficients (LRC, URC) computed as percents from log-transformed data, per Velaquez, et al (J Nucl Med. 2009 Oct;50(10):1646-54. doi: 10.2967/jnumed.109.063347. Epub 2009 Sep 16. PMID: 19759105 ).
  Where Within Subject Coefficient of Variation (wCV) is a percentage defined as wCV(%)=100* (exp( SD[ld]/√2) - 1)
  and LRC and URC are calculated as: RC=100 (exp(±1.96 SD[ld]) -1).
  here SD[ld] is the standard deviation of the difference of the log-transformed PET measurements. These bounds provide an estimate of the lower and upper bounds of percent change observed between scans for each measurement.
Time Frame: Baseline and retest within 1 to 7 days after (but prior to the start of therapy)
Population: Analysis will be performed SUVmax and SUV Peak, average and maximum values, across patients and by target tumor.
Measure: Number (95% Confidence Interval); unit: Within Subj. Coefficient of Variation %
Groups:
- FMISO Reproducibility: Participants with two FMISO PET scans within 1 to 7 days of each other and prior to Visit 2 to test reproducibility of FMISO PET removing 5 participants with protocol variations which could affect the SUV measurements
Arm/Group | FMISO Reproducibility
Number analyzed (Participants) | 29
Within Subj. Coefficient of Variation %
  SUVmax : Average across all lesions by participant | 7.03 [-17.18 to 20.74]
  SUVmax : Maximum across all lesions by participant | 9.60 [-22.43 to 28.92]
  SUVmax : Target Lesion | 8.18 [-19.59 to 24.36]
  SUVpeak: Average across all lesions by participant | 7.08 [-17.27 to 20.88]
  SUVpeak: Maximum across all lesions by participant | 9.20 [-21.65 to 27.63]
  SUVpeak: Target Lesion | 8.24 [-19.71 to 24.55]

4. Secondary Outcome: Correlation Between T/Cmax and T/Bmax
Description: Pearson correlation coefficient will be used to quantify the correlation between T/Bmax, the maximum tissue-to-blood ratio activity value, and T/Cmax, the tissue-to-cerebellum activite value Since T/Cmax does not requiring blood sampling and is image derived, a high correlation would indicate that T/Cmax could be an advantageous surrogate for T/Bmax.
Time Frame: At baseline
Measure: Number; unit: correlation coefficient
Groups:
- DSC MRI: Participant with DSC MRI
Arm/Group | DSC MRI
Number analyzed (Participants) | 38
correlation coefficient | 0.98

5. Secondary Outcome: Correlation Between MRS Markers and MR Imaging Markers of Vascularity as Well as Between MRS Markers and PET Markers of Tumor Hypoxia
Description: Correlation between MRS markers and MR imaging markers and PET markers of tumor hypoxia
  MRS markers include:
  NAA/Cho, Cho/Cr, Lac/Cr, and Lac/NAA measured within tumor and at the periphery.
  MR imaging markers of vascularity include: CBV, CBF, and ktrans PET tumor hypoxia marker: SUVmax
Time Frame: baseline
Population: Seventeen participants from four sites had analyzable 3D MRSI datasets acquired on Philips, GE or Siemens scanners at either 1.5T or 3T. MRSI data were analyzed using LCModel to quantify metabolites N-acetylaspartate (NAA), creatine (Cr), choline (Cho), and lactate (Lac)
Measure: Number; unit: correlation coefficient
Groups:
- nrCBV: 17 participants with measured MRS markers and nRCBV: relative cerebral blood volume, corrected for leakage effects and normalized to normal-appearing white matter;
- nCBF: 17 participants with measured MRS markers and nCBF: cerebral blood flow, normalized to normal-appearing white matter;
- Median K-trans: 17 participants with measured MRS markers and k-trans: vascular permeability
- SUV Max: 17 participants with measured MRS markers and SUVmax: standardized uptake value
Arm/Group | nrCBV | nCBF | Median K-trans | SUV Max
Number analyzed (Participants) | 17 | 17 | 17 | 17
correlation coefficient
  NAA/Cho Tumor | -0.38 | -0.41 | -0.08 | -.33
  NAA/Cho Periphery | -0.33 | -0.34 | 0.14 | -0.41
  Cho/Cr Tumor | 0.24 | 0.28 | -0.2 | 0.03
  Cho/Cr Periphery | 0.17 | 0.20 | -0.27 | 0.11
  Lac/Cr Tumor | -0.27 | -0.25 | -0.06 | -0.29
  Lac/Cr Periphery | -0.09 | -0.11 | 0.10 | -0.15
  Lac/NAA Tumor | -0.02 | -0.01 | 0.23 | -0.18
  Lac/NAA Periphery | -0.01 | -0.01 | 0.33 | -0.04

6. Other Pre Specified Outcome: Overall and Progression Free Survival
Description: Disease progression was defined by Macdonald criteria. Survival and Progression were evaluated every 3months and at the end of study (up to 5 years) and time to event evaluated.
Time Frame: Baseline, every 3 months through study completion (up to 5 years for progression and survivorship)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Newly Diagnosed Glioblastoma Multiforme Patients
Number analyzed (Participants) | 42
days
  Median OS time | 408 [316 to 642]
  Median PFS | 258 [190 to 335]

7. Other Pre Specified Outcome: SUVpeak and T/Bmax as Measures of Tumor Hypoxia
Description: The FMISO image data were normalized by the average blood activity to produce pixel level tissue-to-blood ratio (T/B) values for all image slices. And the severity of the hypoxia was determined by the pixel with the maximum T/B value (TBmax).
  FMISO SUVpeak was determined as the average SUV from a 1 cm circular ROI centered over the hottest pixel. Since FMISO selectively binds to hypoxic tissues, SUVpeak within a region provides a measure of tumor hypoxia.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- FMISO-PET: Quantitative PET measurements Max tumor:blood ratio (TBmax) Peak Standardized uptake Values (SUVpeak)
Arm/Group | FMISO-PET
Number analyzed (Participants) | 38
ratio
  SUVpeak | 2.49 (0.89)
  T/Bmax | 2.13 (0.77)

8. Other Pre Specified Outcome: Hypoxic Volume as a Measure of Tumor Hypoxia
Description: The hypoxic volume (HV) was determined as the volume of pixels in the tumor on in the FMISO\PET with a tumor to blood activity ratio ≥ 1.2.
  HV is a measure of the spatial extent of tumor hypoxia (in milliliters)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | FMISO-PET
Number analyzed (Participants) | 38
milliliters | 14.21 (11.61)

9. Other Pre Specified Outcome: DWI Apparent Diffusion Coefficient (ADC)
Description: Apparent Diffusion Coefficient (ADC) measures water diffusion through tissue (mm^2/s). Cerebral infarction leads to diffusion restriction resulting in a low ADC signal in the infarcted area.
  A double Gaussian mixed model was fit to the ADC histogram and the mean of the lower and the mean of the higher ADC curves were evaluated
Time Frame: baseline
Population: Participants having a usable FMISO\PET and DWI\MRI scans
Measure: Mean (Standard Deviation); unit: mm^2/s
Arm/Group | DWI-MRI
Number analyzed (Participants) | 39
mm^2/s
  Low | 0.99 (0.15)
  High | 1.48 (0.39)

10. Other Pre Specified Outcome: Normalized Relative Cerebral Blood Volume (nRCBV) and Normalized Cerebral Blood Flow (nCBF)
Description: Relative cerebral blood volume (RCBV) maps, computed from the integral of ∆R2*(t), were corrected for leakage effects and normalized to normal appearing white matter (nRCBV); nRCBV provides a measure of tumor vasculature Cerebral blood flow (CBF) maps were was normalized to the mean of the region of interest (ROI) in normal appearing white matter (nCBF); nCBF provides a measure of vascular permeability and perfusion
Time Frame: baseline
Population: Evaluable participants with both usable FMISO\PET and DSC\MRI.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DSC MRI
Number analyzed (Participants) | 37
ratio
  nRCBV | 3.13 (1.86)
  nCBF | 3.36 (2.02)

11. Other Pre Specified Outcome: Summary of Mean and Median Ktrans Across Participants.
Description: ktrans is a measure of vascular permeability and reflects the rate of gadolinium moves from plasma to extravascular extracellular space (predominantly though blood flow and capillary leakage), which can be represented by the mean or median rate.
  Mean & Median ktrans within subject were computed using a matrix-based linearization method to fit tissue ∆R1(t) to the extended Tofts model.
  The mean across subjects is presented below (Mean (Mean-ktrans) and Mean(Median-Ktrans))
Time Frame: baseline
Population: Evaluable patients with usable FMISO\PET and DCE\MRI
Measure: Mean (Standard Deviation); unit: 1/min
Arm/Group | DCE MRI
Number analyzed (Participants) | 31
1/min
  Mean kTrans | 0.04 (0.03)
  Median kTrans | 0.03 (0.07)

ADVERSE EVENTS:
Time Frame: until 24hrs after FMISO administration, evaluated up to 72hours post FMISO injection.
Description: The adverse reporting period is 10 half-lives after the administration of the investigational imaging radiotracer, with a minimum reporting period of at least 24hours post injection. Participants must be reassessed for events between 24 and 72hours post injection.
Groups:
- Evaluable Cases: Patients with Newly diagnosed GBM scheduled to have FMISO PET/CT two weeks before initiation of chemoradiotherapy with temozolomide.
- Diagnostic PET (Using FMISO): Patients with Newly diagnosed GBM who have FMISO PET/CT Imaging two weeks before initiation of chemoradiotherapy with temozolomide.
- Diagnostic MRI (DCE MRI): Patients with Newly diagnosed GBM who have FMISO PET/CT and Dynamic Contrast Enhanced (DCE) MR Imaging two weeks before initiation of chemoradiotherapy with temozolomide.
- Diagnostic MRI (DSE MRI): Patients with Newly diagnosed GBM who have FMISO PET/CT and Dynamic Susceptibility Contrast Enhanced (DSC) MR Imaging two weeks before initiation of chemoradiotherapy with temozolomide.
- Diagnostic MRI (DWI MRI): Patients with Newly diagnosed GBM who have FMISO PET/CT and Diffusion-Weighted Imaging (DWI) MR Imaging two weeks before initiation of chemoradiotherapy with temozolomide.
Arm/Group | Evaluable Cases | Diagnostic PET (Using FMISO) | Diagnostic MRI (DCE MRI) | Diagnostic MRI (DSE MRI) | Diagnostic MRI (DWI MRI)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38 | 0/37 | 0/31 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38 | 0/37 | 0/31 | 0/39
Other Adverse Events (participants affected / at risk) | 0/42 | 0/38 | 0/37 | 0/31 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2012-01-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT00902577/Prot_SAP_ICF_000.pdf